CLINICAL TRIAL: NCT07070284
Title: "Escape 10 Study. Epidemiology and Determinants of Outcomes of Severe Community-acquired Pneumonia in the Elderly"
Brief Title: ESCAPE10: Epidemiology, Risk Factors, and Outcomes of Severe Community-acquired Pneumonia in Elderly PatientsAcquired Pneumonia (sCAP) in Elderly Patients"
Acronym: ESCAPE10
Status: Enrolling by invitation | Type: Observational
Sponsor: Joan Sabater Riera (Other)
Collaborators: European Society of Clinical Microbiology and Infectious Diseases (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Joan Sabater Riera, Head of the Medical Unit, Department of Critical Care, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: ESCAPE10 STUDY
Record Dates: First submitted 2025-06-07; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Severe Community-Acquired Pneumonia (sCAP); Elderly Infection; Community-Acquired Infections; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Community-Acquired Pneumonia; Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Community-Acquired Pneumonia in the Elderly: Participants aged 65 years or older who were hospitalized with radiologically confirmed severe community-acquired pneumonia (sCAP), as defined by protocol criteria. All patients included met clinical and radiological criteria for sCAP and were admitted to an acute care hospital during the defined inclusion period.

SUMMARY:
The ESCAPE 10 study is a multinational, retrospective, observational cohort study that aims to investigate the epidemiology and outcome determinants of severe community-acquired pneumonia (sCAP) in elderly patients (≥65 years). Conducted across multiple European countries, the study will include at least 500 patients admitted to acute care hospitals with radiologically confirmed sCAP, with enrollment distributed evenly between epidemic (winter) and non-epidemic (summer) seasons.

The primary objective is to assess 28-day mortality. Secondary objectives include evaluating in-hospital mortality, pneumonia-related complications, Intensive Care Unit (ICU) stay, ventilation needs, and identifying clinical risk factors associated with poor outcomes. Additionally, the study aims to propose a set of quality indicators for sCAP management and assess gender-related differences and clinical subphenotypes in the post-COVID-19 era.

Data will be retrospectively collected from medical records, with no interventions applied. Findings from this study are expected to guide improvements in clinical care, patient safety, and outcome prediction models in elderly populations with sCAP.

DETAILED DESCRIPTION:
Severe community-acquired pneumonia (sCAP) remains a leading cause of morbidity and mortality in older adults, especially those aged 65 years and above. The ESCAPE 10 study is a multinational, retrospective, observational cohort study designed to explore the epidemiological patterns, clinical characteristics, and outcomes of elderly patients hospitalized with sCAP across diverse European settings.

The study will include at least 500 patients enrolled over a 13-month period (January 1, 2024, to January 31, 2025), with data collection evenly split between epidemic (winter influenza) and non-epidemic (summer) seasons. Participating centers will retrospectively identify eligible patients using standardized inclusion criteria: age ≥65, radiologically confirmed pneumonia, and fulfillment of protocol-defined sCAP criteria. Patients with recent hospitalization, terminal illness, or under palliative care will be excluded.

The primary outcome is 28-day all-cause mortality. Secondary outcomes include in-hospital mortality, pneumonia-attributed mortality, length of hospital and ICU stay, rate of complications (such as Acute Respiratory Distress Syndrome (ARDS), Ventilator-Associated Pneumonia (VAP), septic shock), functional and cognitive status at discharge, and identification of risk factors for adverse outcomes. Quality of care will be assessed through predefined indicators including timeliness of antibiotic administration, adherence to clinical guidelines, and preventive measures like vaccination status.

This study also aims to assess gender differences in sCAP presentation and outcomes, define clinical endotypes, and develop a framework of quality indicators for elderly care in sCAP. No patient interventions will be performed, and data will be extracted from medical records using a secure, coded system Research Electronic Data Capture (REDCap). The results will inform clinical decision-making and quality improvement efforts in the management of sCAP in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years-old or older.
* Patients with clinically and radiologically (Chest X-Ray (CXR), Computerized Tomography (CT) or lung ultrasound (LUS) confirmed pneumonia.
* Patients fulfilling the protocol definition of sCAP

Exclusion Criteria:

* Age < 65 years.
* Recent hospitalization (above 48 h within the past 10 days) in acute healthcare settings.
* Terminal events or imminent death
* Patients receiving comfort care only or with documented decisions to forgo intensive medical interventions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients aged 65 years or older with a clinical and radiological diagnosis of severe community-acquired pneumonia (sCAP). Participants will be enrolled retrospectively from multiple European centers, representing a diverse elderly population. The study includes patients admitted during both epidemic (winter) and non-epidemic (summer) seasons to capture seasonal variations in pathogen distribution and clinical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
28-day All-Cause Mortality | 28 days from admission
  Number of participants who die from any cause within 28 days from the date of hospital admission.

SECONDARY OUTCOMES:
In-Hospital Mortality (All Cause) | From hospital admission through hospital discharge (average of 5 to 30 days)
  Proportion of participants who die from any cause during their hospital stay, from admission to discharge, regardless of length of stay.
Pneumonia-Attributed In-Hospital Mortality | From hospital admission through hospital discharge (average of 5 to 30 days)
  Proportion of participants whose death during hospitalization was determined to be directly attributable to pneumonia, based on physician documentation and medical record review
Length of Hospital Stay (LOS) | Through hospital discharge (average of 5 to 30 days)
  Duration of hospitalization, measured in calendar days from the date of admission to the date of discharge
Duration of ICU Stay | Through ICU or High Dependency Unit (HDU) discharge (average of 2 to 15 days)
  Number of calendar days each participant spends in an Intensive Care Unit (ICU) or High-Dependency Unit (HDU), from ICU/HDU admission to ICU/HDU discharge.
Duration of Mechanical Ventilation | Through hospital discharge (average of 2 to 20 days)
  Total number of calendar days a participant receives invasive or non-invasive mechanical ventilation during hospitalization.
Rate of Pneumonia-Related Complications | From hospital admission to hospital discharge, up to a maximum of 30 days
  Incidence of complications such as ARDS, septic shock, bacteremia, empyema, or VAP
Functional Status at Discharge | At hospital discharge (typically between Day 5 and Day 30 post-admission, depending on clinical course)
  Assessment of the patient's physical functional level at the time of hospital discharge, using standardized scales such as the Barthel Index or Clinical Frailty Scale, when available. The chosen scale will be specified in each case.
  Units of Measure: Score on a standardized functional scale (e.g., Barthel Index, 0-100, where higher scores indicate better function; or Clinical Frailty Scale, 1-9, where higher scores indicate worse function)
Cognitive Function at Discharge | At hospital discharge (typically between Day 5 and Day 30 post-admission, depending on clinical course)
  Evaluation of cognitive status at the time of hospital discharge using available documentation from the medical record and/or validated tools such as the Confusion Assessment Method (CAM) or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) when available. Presence or absence of delirium and/or cognitive decline will be recorded.
  Units of Measure: Cognitive function status (e.g., presence or absence of delirium based on CAM or CAM-ICU; categorical assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rello, phD, MD, Principal Investigator — European Study Group Infections in the Elderly. ESCMID
Locations (18):
- University Hospital for Infectious Diseases Dr. Fran Mihaljević, Zagreb, City of Zagreb, Croatia
- France (5):
  - Thibaut Fraisse, Alès
  - Centre Hospitalier Intercommunal Hôpitaux du Pays du Mont-Blanc - Site de Chamonix, Chamonix
  - Centre hospitalier Alpes Léman, Contamine-sur-Arve
  - Centre Hospitalier de Melun, Melun
  - Hôpital Bichat - Claude-Bernard, Paris
- Evangelismos General Hospital, Athens, Greece
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome, Lazio
  - ASST del Garda - Ospedale Civile "La Memoria" di Gavardo, Gavardo, Lombardy
  - ARNAS Civico-Di Cristina-Benfratelli Hospital - Infectious Diseases Unit, Palermo, Sicily
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, Tuscany
- Centro Hospitalar Universitário de São João (CHUSJ), Porto, Portugal
- Spain (5):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Bellvitge Universitary Hospital, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar Barcelona, Barcelona, Catalonia
  - Corporació Sanitària Parc Taulí, Sabadell, Catalunuya
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT07070284/Prot_SAP_000.pdf